CLINICAL TRIAL: NCT05005429
Title: A Phase II Single Arm Clinical Trial Assessing the Efficacy and Safety of BIntrafusp Alfa (M7824) in Previously Treated Advanced Malignant Pleural MESothelioma (BIMES)
Brief Title: Study of the Efficacy and Safety of the Bintrafusp Alfa in Previously Treated Advanced Malignant Pleural Mesothelioma
Acronym: BIMES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 20/09_BIMES; 2020-004902-67 (EudraCT Number)
Record Dates: First submitted 2021-08-10; First posted 2021-08-13 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Mesothelioma; Lung
Keywords: Malignant pleural mesothelioma; Bintrafusp alfa
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Bintrafusp alfa (M7824) (Experimental): Bintrafusp alfa (M7824): 1200mg, over 60 minutes IV infusion The treatment will start within 1-5 days from enrollment. The treatment will be administered at day 1 of 14-day intervals .
  Treatment will be administered until unacceptable toxicity, loss of clinical benefit, disease progression or completion of 2 years of therapy. If the patient has benefit after 2 years, the trial chair and the sponsor must be consulted to evaluate how to continue with the treatment.
  Interventions: Drug: Bintrafusp alfa

INTERVENTIONS:
Drug: Bintrafusp alfa — Bintrafusp alfa (M7824) is a bifunctional fusion protein composed of the extracellular domain of the transforming growth factor β (TGF-β) receptor II (a TGF-β "trap") fused to a human immunoglobulin G1 antibody blocking programmed death-ligand 1 (PD-L1).
  Day 1 of week 1 of treatment will start within 1-5 days from enrollment. Cycles will be administered every 2 weeks (±3 days) until progression or other reason to discontinue. If a pseudoprogression is suspected patient is allowed to continue treatment until loss of clinical benefit as judged by principal investigator and after the permission from the trial chair is granted.
  On Day 1 of each cycle (QW2), all eligible patients will receive:
  Bintrafusp alfa (M7824): 1200mg, IV infusion over 60 minutes Current experience revealed that IRRs to bintrafusp alfa occur seldomly and are generally mild to moderate in severity. Therefore, administration of a premedication is generally not required.
  Other Names: M7824

SUMMARY:
This is an open-label, non-randomized, phase II, single arm, multi-center controlled clinical trial.

47 patients will be enrolled in this trial to determine the efficacy and safety of Bintrafusp alfa (M7824) in advanced malignant pleural mesothelioma patients previously treated with platinum-based chemotherapy.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, phase II, single arm, multi-center controlled clinical trial.

Patients enrolled will receive Bintrafusp alfa (M7824) 1200mg intravenous. The treatment will be administered at day 1 of 14-day intervals.Treatment will be administered until unacceptable toxicity, loss of clinical benefit, disease progression or completion of 2 years of therapy.

The primary objective is to determine the efficacy of M7824 in terms of the Progression Free Survival (PFS) assessed by the investigator according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST) Version 1.1.

Patient accrual is expected to be completed within 1.5 years excluding a run-in-period of 3-6 months. Treatment and follow-up are expected to extend the study duration to a total of 3.5 years. Patients will be followed 1 month after treatment. The study will end once survival follow-up has concluded.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 18 years and capable of giving signed informed consent or requirement per local legislation.
* ECOG performance status of 0-2.
* Histologically confirmed malignant pleural mesothelioma (all histological subtypes are eligible), unresectable advanced or metastatic.
* Patients that progressed or be intolerant to ≤ 2 regimens of chemotherapy, including platinum-based chemotherapy with pemetrexed. Prior bevacizumab treatment given during chemotherapy are allowed.
* Evaluable disease or measurable disease as assessed according to the modified RECIST v1.1 criteria.
* Availability of tumor tissue for translational research (at least 10 slides); Archival tumor tissue at diagnosis can be sent if it was obtained less than 18 months ago.
* Life expectancy of at least 3 months.
* Adequate hematologic and organ function defined by the following laboratory results obtained within 14 days prior to enrollment:

Hematologic: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL Hepatic: Total bilirubin level ≤ the upper limit of normal (UNL) range, AST and ALT levels ≤ 1.5 x ULN and ALP ≤ 2.5 x ULN. For participants with liver involvement in their tumor, AST ≤5 x ULN, ALT ≤ 5 x ULN, and bilirubin ≤ 3.0 x ULN.

Renal: Creatinine level ≤1.5 x ULN or estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method) For participants with Creatinine > 1.5 x ULN, glomerular filtration rate (GFR) can also be used.

Coagulation: normal international normalized ratio (INR), PT ≤ 1.5 x ULN and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN.

* Stable HIV infection on ART for at least 4 weeks, no documented evidence of multi-drug resistance, viral load of < 400 copies/ml and CD4+ T-cells ≥ 350 cells/μL.
* Controlled HBV/HCV infection on a stable dose of antiviral therapy, HBV viral load below the limit of quantification. HCV viral load below the limit of quantification.
* All patients are notified of the investigational nature of this study and signed a written informed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention.
* For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly throughout the study and for at least 2 months after last bintrafusp alfa treatment administration .
* For male patients with female partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate [< 1% per year] when used consistently and correctly.
* Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 8 days prior to initiation of study drug.

Exclusion Criteria:

* Prior immune checkpoint therapy with an anti-PD-1, anti-PD-L1, anti-CD137, or anti-CTLA-4 antibody.
* Known severe hypersensitivity [Grade ≥ 3 NCI CTCAE 5.0]) to investigational product or any component in its formulations, any history of anaphylaxis, or recent, within 5 months, history of uncontrollable asthma.
* Previous malignant disease (other than the target malignancy to be investigated in this study) within the last 3 years. Participants with a history of cervical carcinoma in situ, superficial or noninvasive bladder cancer, localized prostate cancer or basal cell or squamous cell carcinoma in situ previously treated with curative intent and endoscopically resected GI cancers limited to the mucosal layer without recurrence in > 1 year are NOT excluded.
* Active central nervous system (CNS) metastases and/or carcinomatous meningitis that require therapeutic intervention or are causing clinical symptoms. Patients with previously treated brain metastases may participate provided the participants are stable and are not using steroids for at least 7 days prior to randomization.
* Prior major surgery within 4 weeks prior to the first dose of study intervention.
* Unstable or unresolved surgical or chemotherapy-related toxicity that would compromise the patient's capacity to participate in the trial. Persisting Grade > 1 NCI CTCAE 5.0 toxicity (except alopecia and vitiligo) related to prior therapy; however, sensory neuropathy Grade ≤ 2 is acceptable.
* Prior organ transplantation including allogenic stem-cell transplantation, except transplants that do not require immunosuppression.
* Live vaccines given 30 days prior to first dose of protocol treatment (M7824). Seasonal flu vaccines that do not contain a live virus are permitted. Also, COVID-19 vaccines approved by the authorities that do not contain live virus are permitted.
* Drug-induced interstitial lung disease (ILD) or participant has had a history of drug-induced pneumonitis that has required oral or IV steroids, and/or other diseases, which in the opinion of the Investigator might impair the participant's tolerance for the study or ability to consistently participate in study procedures.
* Active and serious autoimmune disease that might deteriorate upon treatment with immunotherapy. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible. Replacement therapy (i.e. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) or topical therapy (e.g., steroids) for psoriasis or eczema is not considered a form of systemic treatment.
* Ongoing clinically serious infections requiring systemic antibiotic or antiviral, antimicrobial, or antifungal therapy.
* Known history of active tuberculosis or any active infection requiring systemic therapy.
* Patients with diagnosed immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to randomization.
* Clinically significant cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* History of bleeding diathesis or recent major bleeding events (i.e. Grade ≥ 2 bleeding events in the month prior treatment)
* Patients with any serious underlying medical condition that might impair patient's capacity to participate in the trial.
* Substance or alcohol abuse, medical, psychological or social conditions that may interfere with the patient's participation in the trial or evaluation of the trial results.
* Women who are pregnant or in the period of lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Principal Investigator — Fundación GECP President
Locations (15):
- Spain (15):
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona, Barcelona
  - Hospital Parc Taulí, Barcelona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Basurto, Bilbao, Bilbao
  - ICO Girona, Hospital Josep Trueta, Girona, Girona
  - Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Virgen De La Victoria, Málaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo, Oviedo
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: Bintrafusp Alfa (M7824)
Started | 47
Completed | 46
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: 47 patients were enrolled in the study although patient 05000013 was finally considered as inclusion error and did not enter in the analysis.
Arm/Group | Experimental: Bintrafusp Alfa (M7824)
Number analyzed (Participants) | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 36
Age, Continuous [Mean (Full Range); unit: years] | 70 [41 to 84]
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 45
  Latin | 1
Smoking habit [Count of Participants; unit: Participants]
  Never smoker (<= 100 cigarettes/lifetime) | 18
  Former smoker (>= 1 year) | 22
  Active smoker | 6
Lines of therapy [Count of Participants; unit: Participants]
  Second (received at least 1 previous line) | 39
  Third (received two previous lines) | 7

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Efficacy of the Treatment
Description: To determine the efficacy of M7824 in terms of the Progression Free Survival (PFS) assessed by the investigator according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST) Version 1.1. Progression is defined using Response Evaluation Criteria in Solid Tumors (mRECIST) Version 1.1 as an increase of at least 20%in the sumof thediameters of viable (enhancing) target lesions, taking as reference the smallest sumof thediameters of the viable (enhancing) target lesions. The sum must also demonstrate an absoluteincrease of at least 5 mm.
Time Frame: From administration of first dose of bintrafusp alfa until objective tumor progression or death, up to 2 years.
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Months
Arm/Group | Experimental: Bintrafusp Alfa (M7824)
Number analyzed (Participants) | 46
Months | 1.9 [1.7 to 5.4]

ADVERSE EVENTS:
Time Frame: Adverse events must be recorded and followed from the day patient signs the Informed consent for the study to 30 days from last dose of administration, up to 2 years.
Arm/Group | Experimental: Bintrafusp Alfa (M7824)
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 22/46
Other Adverse Events (participants affected / at risk) | 16/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Bintrafusp Alfa (M7824) (N=46)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2)
Allergic reaction (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 9 (9)
Colitis (Gastrointestinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Oher (Skin and subcutaneous tissue disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Bintrafusp Alfa (M7824) (N=46)
Adrenal Insufficiency (Endocrine disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No study limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT05005429/Prot_SAP_000.pdf